CLINICAL TRIAL: NCT03407638
Title: PRimary Care Opioid Use Disorders Treatment (PROUD) Trial
Acronym: PROUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CTN-0074; UG1DA040314 (NIH)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder
Keywords: Opioid Use Disorder; Primary Care; Buprenorphine; Naltrexone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Pragmatic Trial: Six health systems are participating in a pragmatic, cluster-randomized, quality improvement trial (hybrid Type III implementation trial). Each of the 6 health systems provided 2 PC clinics willing to be in the randomized controlled trial. Each health system will implement collaborative care for OUD treatment in one randomly selected PC clinic. All data used to evaluate primary and secondary outcomes are secondary data from the EHR or insurance claims.
Masking Description: Statistical analysts (biostatisticians) who analyze trial results will be masked for objectives 1 and 2.
  Main analyses of the primary outcome will be conducted by the National Drug Abuse Treatment Clinical Trials Network (NDAT CTN) Data and Statistics Center (DSC). The de-identified dataset provided to the DSC by the data management team at Kaiser Permanente Washington Health Research Institute will have the identity of the intervention and Usual Primary Care clinic at each site masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROUD Intervention (Active Comparator): Primary care clinics randomized to the PROUD Intervention will implement the Massachusetts (MA) Model of collaborative care for opioids use disorders (OUDs). The PROUD trial provides financial support to cover the nurse case manager (NCM) salary and technical assistance for the duration of the study, but the health systems-not investigators-implement the MA Model as part of quality improvement, and the health system and its clinicians provide all clinical care.
  Interventions: Other: PROUD Intervention
- Usual Primary Care (No Intervention): Clinics randomized to usual primary care do not receive any resources or support from the study but are free to improve opioid use disorder (OUD) care in any way they choose.

INTERVENTIONS:
Other: PROUD Intervention — The PROUD intervention includes 3 strategies used to implement the MA Model: 1. Clinic leadership receives funding for a 1.0 full time equivalent NCM for 2 years after randomization and technical support for recruiting and hiring the NCM. Once hired for the study, the NCM will receive technical assistance (TA) from experts at Boston Medical Center (BMC) supported by PROUD, but NCMs will be employed and supervised by the health system. 2. Experts at BMC who originally developed and disseminated the MA Model will: provide intervention clinics with a Manual; train PROUD NCMs at BMC; and provide the ongoing TA for 2 years after randomization. 3. At least 3 primary care providers in the PROUD intervention clinic will obtain DEA waivers to prescribe buprenorphine for OUDs, if not already waivered, and work closely with the NCM to offer high quality primary care for OUDs (e.g. medication treatment with buprenorphine or naltrexone with close follow-up to maximize retention in treatment).
  Arms: PROUD Intervention

SUMMARY:
Effective treatment for opioid use disorders (OUDs) requires medications. Two medications for treating OUDs-buprenorphine and injectable naltrexone-can be prescribed in primary care (PC). However, despite the current opioid epidemic and expert recommendations that OUDs should be treated in PC, most PC clinics do not offer treatment for OUDs. This reflects a lack of consensus among health system leaders and clinicians that OUDs should be treated in PC.

The PRimary care Opioid Use Disorders treatment (PROUD) Trial is a pragmatic cluster-randomized, quality improvement trial that evaluates implementation of a team-based approach to PC supported by a full time nurse (the "PROUD intervention"). This type of team-based PC is often referred to as "collaborative care" for management of OUDs in PC, and this type of trial is often referred to as a Hybrid Type III implementation trial.

The trial is being conducted in 6 diverse health systems spanning 5 states (New York, Florida, Michigan, Texas, and Washington), with 2 PC clinics in each system randomized. One clinic is randomly selected to implement the PROUD intervention and the other continues usual PC (UPC).

The overall objective of the PROUD trial is to provide information to guide health system leaders who are faced with the decision of whether or not to treat OUDs in PC, by evaluating the benefits of implementing the PROUD intervention that integrates high quality OUD treatment (i.e. buprenorphine or injectable naltrexone) into the normal flow of PC.

The primary objective of the PROUD trial is to evaluate whether the PROUD intervention increases OUD treatment with buprenorphine or injectable naltrexone, documented in the electronic health records (EHRs) of PC patients, over a 2 year follow-up, as compared to UPC.

The primary hypothesis is that there will be a significant increase in the number of patient-days of medication treatment for OUDs documented in the EHR of PC patients in the 2 years after clinics are randomized to the PROUD intervention compared to PC clinics randomized to UPC. This implementation objective reflects whether the PROUD intervention increases initiation of and/or retention in OUD treatment, documented in EHRs within medical settings.

The main secondary objective is to test the hypothesis that PC patients with OUDs documented in their EHRs in the 3 years prior to randomization who receive care in PROUD intervention clinics, compared to those who receive care in UPC clinics, will have fewer days of acute care utilization (including urgent care, emergency department [ED] and hospital care) in the 2 years after randomization. This effectiveness objective assesses whether implementation of the MA Model improves patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The 12 clinics were eligible if their health system leaders agreed they would participate prior to study start.

Patients are eligible for inclusion in the sample for analyses of the PROUD trial if they visited one of the randomized clinics at any time in the 5 year study period. Specific inclusion criteria for the trial are:

1. Age is 16 to 90 years at any time during the study; and
2. Visited a PROUD trial primary care clinic in the 3 years prior to randomization or the 2 years after (note: one of the 6 study sites may only be able to provide EHR data for 2 years before randomization)

Exclusion Criteria:

* Patients who have requested through their health systems to opt out of research will be excluded from this study.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 973759 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Patient-days of OUD medication treatment | 2-year period post-randomization
  Clinic-level number of patient-days of OUD treatment with buprenorphine and injectable naltrexone documented in the EHR during the period from randomization until two years after, reported per 10,000 primary care patients in the clinic in the 2 years post-randomization (reported as patient-years of treatment per 10,000).

SECONDARY OUTCOMES:
Acute care utilization | 2-year period post-randomization
  Patient-level number of days of acute care utilization during the period from randomization until two years after, among patients with an OUD diagnosis documented in the EHR in the three years prior to randomization.

OTHER OUTCOMES:
Newly recognized OUDs | 2 years after randomization
  Clinic-level number of patients with a new International Classification of Disease (ICD) code for OUD documented in the EHR during the period from randomization until two years after who did not have an OUD diagnosis documented in the EHR in the two years prior to randomization, reported per 10,000 primary care patients in the clinic in the 2 years post-randomization.
Initiation of OUD treatment | 2 years after randomization
  Clinic-level number of patients who initiate (1) buprenorphine or (2) injectable naltrexone with an OUD diagnosis as documented in the EHR during the period from randomization until two years after, reported per 10,000 primary care patients in the clinic in the 2 years post-randomization. Measure will be calculated for any initiation.
Retention in OUD treatment | 2 years after randomization
  Clinic-level number of patients with OUD treatment during the period from randomization until two years after randomization as documented in the EHR, who also receive OUD treatment on 80% of days available after initiation, reported per 10,000 primary care patients in the clinic in the 2 years post-randomization.
Urgent care or ED use | 2 years after randomization
  Patient-level number of visits to urgent care or EDs during the period from randomization until two years after, among patients with an OUD diagnosis documented in the EHR in the three years prior to randomization.
Inpatient Days hospitalized | 2 years after randomization
  Patient-level number of days hospitalized during the period from randomization until two years after, among patients with an OUD diagnosis documented in the EHR in the three years prior to randomization.
Naloxone prescribing | 2 years after randomization
  Patient-level number of prescriptions of naloxone for overdose management in the period from randomization until two years after, among patients with an OUD diagnoses in the three years prior to randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine A Bradley, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (6):
- United States (6):
  - University of Miami Health System, Miami, Florida
  - Henry Ford Health System, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Harris Health System, Houston, Texas
  - Kaiser Permanente Washington, Seattle, Washington
  - MultiCare Health System, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
The NIDA Data Share website will include a description of the PROUD trial's main analytic dataset supporting the primary objective and information on how to obtain the dataset, which must remain de-identified. Investigators wishing to obtain PROUD study data should contact the Lead Investigator to discuss the dataset request. Requests will be reviewed on a case-by-case basis and may require funding to support 1) programming to create the necessary de-identified analytic dataset(s) and 2) establish a data transfer agreement and IRB approval. The NIDA Data Share website will explicitly indicate that data elements for site or clinic may be obtained, but access will be highly restricted and will need the appropriate agreements and approvals in place. If data on sites and clinics are provided, names will be masked. De-identification includes masking all dates and zip codes prior to providing the data.
Supporting Information: Study Protocol, SAP
Time Frame: Investigators will review requests at any time now that the primary paper is published.
Access Criteria: Sharing of de-identified datasets will be determined on a case-by-case basis by the Lead Investigator.
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Background] Alford DP, LaBelle CT, Kretsch N, Bergeron A, Winter M, Botticelli M, Samet JH. Collaborative care of opioid-addicted patients in primary care using buprenorphine: five-year experience. Arch Intern Med. 2011 Mar 14;171(5):425-31. doi: 10.1001/archinternmed.2010.541. PMID 21403039
- [Background] LaBelle CT, Han SC, Bergeron A, Samet JH. Office-Based Opioid Treatment with Buprenorphine (OBOT-B): Statewide Implementation of the Massachusetts Collaborative Care Model in Community Health Centers. J Subst Abuse Treat. 2016 Jan;60:6-13. doi: 10.1016/j.jsat.2015.06.010. Epub 2015 Jun 26. PMID 26233698
- [Derived] Lapham GT, Hyun N, Bobb JF, Wartko PD, Matthews AG, Yu O, McCormack J, Lee AK, Liu DS, Samet JH, Zare-Mehrjerdi M, Braciszewski JM, Murphy MT, Arnsten JH, Horigian V, Caldeiro RM, Addis M, Bradley KA. Nurse Care Management of Opioid Use Disorder Treatment After 3 Years: A Secondary Analysis of the PROUD Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2447447. doi: 10.1001/jamanetworkopen.2024.47447. PMID 39576637
- [Derived] Bobb JF, Idu AE, Qiu H, Yu O, Boudreau DM, Wartko PD, Matthews AG, McCormack J, Lee AK, Campbell CI, Saxon AJ, Liu DS, Altschuler A, Samet JH, Northrup TF, Braciszewski JM, Murphy MT, Arnsten JH, Cunningham CO, Horigian VE, Szapocznik J, Glass JE, Caldeiro RM, Tsui JI, Burganowski RP, Weinstein ZM, Murphy SM, Hyun N, Bradley KA. Offering nurse care management for opioid use disorder in primary care: Impact on emergency and hospital utilization in a cluster-randomized implementation trial. Drug Alcohol Depend. 2024 Aug 1;261:111350. doi: 10.1016/j.drugalcdep.2024.111350. Epub 2024 Jun 10. PMID 38875880
- [Derived] Wartko PD, Bobb JF, Boudreau DM, Matthews AG, McCormack J, Lee AK, Qiu H, Yu O, Hyun N, Idu AE, Campbell CI, Saxon AJ, Liu DS, Altschuler A, Samet JH, Labelle CT, Zare-Mehrjerdi M, Stotts AL, Braciszewski JM, Murphy MT, Dryden D, Arnsten JH, Cunningham CO, Horigian VE, Szapocznik J, Glass JE, Caldeiro RM, Phillips RC, Shea M, Bart G, Schwartz RP, McNeely J, Liebschutz JM, Tsui JI, Merrill JO, Lapham GT, Addis M, Bradley KA; PROUD Trial Collaborators; Ghiroli MM, Hamilton LK, Hu Y, LaHue JS, Loree AM, Murphy SM, Northrup TF, Shmueli-Blumberg D, Silva AJ, Weinstein ZM, Wong MT, Burganowski RP. Nurse Care Management for Opioid Use Disorder Treatment: The PROUD Cluster Randomized Clinical Trial. JAMA Intern Med. 2023 Dec 1;183(12):1343-1354. doi: 10.1001/jamainternmed.2023.5701. PMID 37902748
- [Derived] Campbell CI, Saxon AJ, Boudreau DM, Wartko PD, Bobb JF, Lee AK, Matthews AG, McCormack J, Liu DS, Addis M, Altschuler A, Samet JH, LaBelle CT, Arnsten J, Caldeiro RM, Borst DT, Stotts AL, Braciszewski JM, Szapocznik J, Bart G, Schwartz RP, McNeely J, Liebschutz JM, Tsui JI, Merrill JO, Glass JE, Lapham GT, Murphy SM, Weinstein ZM, Yarborough BJH, Bradley KA. PRimary Care Opioid Use Disorders treatment (PROUD) trial protocol: a pragmatic, cluster-randomized implementation trial in primary care for opioid use disorder treatment. Addict Sci Clin Pract. 2021 Jan 31;16(1):9. doi: 10.1186/s13722-021-00218-w. PMID 33517894
- [Derived] Bobb JF, Qiu H, Matthews AG, McCormack J, Bradley KA. Addressing identification bias in the design and analysis of cluster-randomized pragmatic trials: a case study. Trials. 2020 Mar 23;21(1):289. doi: 10.1186/s13063-020-4148-z. PMID 32293514